CLINICAL TRIAL: NCT01465711
Title: Diagnostic Accuracy of Pancreatic Stone Protein in Predicting Severe Outcome in Patients With Peritonitis at the Intensive Care Unit
Brief Title: The Value of PSP in Predicting Outcome in ICU Surgical Peritonitis Patients
Status: Completed | Type: Observational
Sponsor: University of Magdeburg (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Antje Wiede, Investigator, University of Magdeburg
Other Study IDs: 33/01
Record Dates: First submitted 2011-10-28; First posted 2011-11-07 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2011-11

CONDITIONS: Peritonitis; Sepsis; Multiple Organ Failure; Death
Keywords: Peritonitis; Sepsis; General Surgery; Intensive Care Units; Sensitivity and Specificity
MeSH Terms: conditions — Peritonitis; Sepsis; Multiple Organ Failure; Death; Hypersensitivity | interventions — Surgical Procedures, Operative; Intubation; Intubation, Intratracheal; Tracheostomy; X-Rays

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum, plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: Admission to the Intensive Care Unit (ICU) after abdominal surgery without suspicion / evidence of peritonitis.
  Interventions: Procedure: All abdominal surgical procedures; Procedure: Intubation; Radiation: Imaging
- Peritonitis: Admission to the Intensive Care Unit (ICU) after abdominal surgery with suspicion / evidence of peritonitis
  Interventions: Procedure: All abdominal surgical procedures; Procedure: Intubation; Radiation: Imaging

INTERVENTIONS:
Procedure: All abdominal surgical procedures — Laparotomy, Laparoscopy
  Other Names: surgical procedures
Procedure: Intubation — Ventilatory support
  Other Names: Endotracheal Intubation, tracheostomy
Radiation: Imaging — Abdominal ultrasound Computer Tomography Magnetic Resonance Imaging
  Other Names: Any type of diagnostic or interventional imaging technique

SUMMARY:
The purpose of this study is to determine the diagnostic accuracy of Pancreatic Stone Protein (PSP) in predicting patient outcomes with suspected peritonitis in the Intensive Care Unit after abdominal surgery and compare PPS with other blood parameters, including C-Reactive Protein (CRP), White Cell Count (WCC), Interleucin-6 (IL-6) and Procalcitonin (PCT).

DETAILED DESCRIPTION:
Peritonitis is a severe complication after abdominal surgery. Patients admitted at the Intensive Care Unit (ICU) following surgery bear the risk of localized infection, sepsis or septic shock. Prevention or early detection of such events is important to intervene with an appropriate therapeutic action and avoid risking a potentially life-threatening situation. White blood cell counts (WCC) and C-Reactive Protein (CRP), Interleucin-6 (IL-6) and Procalcitonin (PCT) have all been promising parameters, however, they are useful only in selective cases and have a limited diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal surgery.
* Admission to the Intensive Care Unit (ICU).
* Blood sampling within 3 hours from admission to the ICU
* Patient over 18 years of age

Exclusion Criteria:

* Patients already treated for peritonitis.
* Patients referred from other hospitals with suspicion of peritonitis
* Patient age less than 18 years of age.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2007-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Localization of Peritonitis | up to 2 months
  Localised vs. diffused. A clinical finding intra-operatively and/or radiologically (i.e. CT or MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Halangk, PhD, Principal Investigator — University of Magdeburg, Department of General, Visceral and Vascular Surgery, Leipziger Str. 44, DE-39120, Magdeburg, Germany; Hans-Ulrich Schulz, MD, Principal Investigator — University of Magdeburg, Department of General, Visceral and Vascular Surgery, Leipziger Str. 44, DE-39120, Magdeburg, Germany; Rolf Graf, PhD, Principal Investigator — University Hospital Zurich, Department of Surgery, Raemistrasse 100, CH-8091, Zurich, Switzerland
Locations (1):
- University of Magdeburg, Magdeburg, Germany

REFERENCES:
- [Derived] Gukasjan R, Raptis DA, Schulz HU, Halangk W, Graf R. Pancreatic stone protein predicts outcome in patients with peritonitis in the ICU. Crit Care Med. 2013 Apr;41(4):1027-36. doi: 10.1097/CCM.0b013e3182771193. PMID 23399938